CLINICAL TRIAL: NCT00601913
Title: CCCWFU 60307 - Pilot Study to Evaluate the Anti-tumor Effect of Erlotnib Administered Befor Surgery in Operable Patients With Squamous Cell Carcinoma of the Head and Neck (HNSCC)
Brief Title: Erlotinib and Surgery in Treating Patients With Head and Neck Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00004038; P30CA012197 (NIH); CCCWFU-60307 (Other: Comprehensive Cancer Center of WFUHS); NCT01588613 (obsolete NCT alias)
Record Dates: First submitted 2008-01-24; First posted 2008-01-28 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage I verrucous carcinoma of the larynx; stage I verrucous carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride; Blotting, Western; Immunohistochemistry; Chromatography, Liquid; Mass Spectrometry; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erlotinib (Experimental): Erlotinib
  Interventions: Drug: erlotinib hydrochloride; Genetic: protein analysis; Genetic: western blotting; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: liquid chromatography; Other: mass spectrometry; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: erlotinib hydrochloride
Genetic: protein analysis
Genetic: western blotting
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: liquid chromatography
Other: mass spectrometry
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment with erlotinib.

PURPOSE: This clinical trial is studying how well erlotinib works when given before surgery in treating patients with head and neck cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify tissue biomarkers (primarily the level of phosphorylation of individual C-terminal EGFR tyrosine sites, measured by nano-LC-MS/MS and markers of main downstream pathways activation such as P-AKT and P-ERK, measured by nano-LC-MS/MS and by more clinically standardized IHC) that best associate with response to neoadjuvant erlotinib hydrochloride treatment in patients with resectable squamous cell carcinoma of the head and neck (HNSCC).
* Determine the best correlations between levels and changes of different individual biomarkers (e.g., levels of C-terminal EGFR phosphorylation and recruited adaptors and markers of downstream pathways activation) in order to evaluate the mechanisms of EGFR pathway activation in HNSCC and mechanisms of EGFR pathway inhibition by erlotinib hydrochloride in HNSCC tissue.
* Evaluate post-erlotinib hydrochloride up-regulation of different receptors and molecules such as HER2 and 3, PDGFR, IGFR, mTOR, src, and aurora kinases, for which there are already specific inhibitors available for clinical studies.

Secondary

* Evaluate the efficacy by overall response, safety, and tolerability of erlotinib hydrochloride before surgery in these patients.
* Evaluate the role of FDG-PET scan as a predictor of response to erlotinib hydrochloride.
* Evaluate the role of PET/CT in measuring the response to short-term treatment with erlotinib hydrochloride.
* Evaluate incidence of risk factors for relapse in the surgical pathology specimens.

OUTLINE: Patients are grouped according to smoking status (non-actively smoking [not smoking, smoking an average of < 10 cigarettes daily, or smoking for < 1 year prior to enrollment] vs actively smoking [smoking an average of ≥ 10 cigarettes daily and smoking for ≥ 1 year]).

* Non-actively smoking patients: Patients receive oral erlotinib hydrochloride 150 mg once daily for at least 14 days. At day 15 patients undergo surgical resection of the tumor.
* Actively smoking patients: Patients receive oral erlotinib hydrochloride 300 mg once daily for at least 14 days. At day 15 patients undergo surgical resection of the tumor.

Patients undergo biopsies at baseline and after completion of study treatment. Tissue samples are analyzed by nano-liquid chromatography and mass spectrometry (nano-LC-MS/MS) for markers of activation and inhibition of different EGFR downstream pathways: PKC, c-Cbl, P-Erk, P- Akt, P-RAF, src, STAT3 and 5, cyclin D1, and D3, p21 and p27, c-fos, E-cadherin, vimentin, and correlative up-regulated receptors: Her 2, Her 3, Cox-2, IGF, VEGF, PDGFR, or other kinases such as src and aurora kinases A and B. The results are confirmed by western blot, protein array, and immunohistochemistry.

After completion of study treatment, patients are followed at 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma (SCC) of the oral cavity, oropharynx, hypopharynx, or larynx

  * SCC of the base of the tongue, pharynx, larynx, or hypopharynx are eligible provided additional biopsy tissue has been already saved in the Tumor Tissue Core Laboratory for research purposes
  * SCC of the oral cavity or tonsils are eligible only if they already have or agree to have additional biopsies of tumor with adjacent normal tissue available for molecular studies
* Candidate for surgical treatment with an established date for surgery with ≥ a 15 day window of opportunity
* Measurable disease by CT scan or MRI
* No nasopharyngeal carcinoma

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* ANC > 1,500/µL
* Platelet count > 100,000/µL
* Total bilirubin < 1.5 mg/dL
* AST/ALT < 2 times upper limit of normal
* Creatinine < 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
  * Significant history of uncontrolled cardiac disease (i.e., uncontrolled hypertension, unstable angina, or myocardial infarction within the past 3 months)
  * Uncontrolled congestive heart failure
  * Cardiomyopathy with decreased ejection fraction
* History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on chest CT scan
* Clinically significant ophthalmologic abnormalities
* HIV positivity

PRIOR CONCURRENT THERAPY:

* More than 1 year since prior chemotherapy, biologic therapy, or hormonal therapy
* No prior radiotherapy or chemotherapy for this tumor
* No prior EGFR inhibitors
* No concurrent grapefruit or grapefruit juice
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Identify tissue biomarkers of EGFR activation and inhibition for which initial values and changes after treatment with erlotinib hydrochloride would best correlate with the objective response of the tumor measured clinically and radiologically

SECONDARY OUTCOMES:
Objective response
Tumor cell metabolic response measured by PET scan at 4-6 days after beginning of treatment and correlation with tumor response evaluated at the end of treatment by CT scan, PET scan, and direct tumor measurements
Role of PET/CT scan in evaluating response to short-term treatment with erlotinib hydrochloride and comparison with the same response evaluation performed by CT scan
Incidence of risk factors for relapse
Incidence of adverse effects or significant laboratory changes
Any treatment-induced delay of the established date for definitive surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Porosnicu, MD, Principal Investigator — Wake Forest University Health Sciences; J. D. Browne, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Porosnicu M, O'Brien Cox A, Waltonen JD, Bunch PM, D'Agostino R, Lycan TW, Taylor R, Williams DW 3rd, Chen X, Shukla K, Kouri BE, Walker T, Kucera G, Patwa HS, Sullivan CA, Browne JD, Furdui CM. Early [18]FDG PET/CT scan predicts tumor response in head and neck squamous cell cancer patients treated with erlotinib adjusted per smoking status. Front Oncol. 2022 Aug 30;12:939118. doi: 10.3389/fonc.2022.939118. eCollection 2022. PMID 36110959